CLINICAL TRIAL: NCT05738057
Title: Combined Therapy Using D-TACE, Gemcitabine and Cisplatin Chemotherapy, and PD1 Antibody for Patients With Advanced and Unresectable Intrahepatic Cholangiocarcinoma: a Single-center, Single-arm Trial
Brief Title: Combined Therapy Using D-TACE, Gemcitabine and Cisplatin, and PD1 Antibody in Advanced and Unresectable Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hua Li (Other)
Responsible Party: Sponsor-Investigator, Hua Li, Director, Hepatic Surgery Department of Third Affiliated Hospital, Sun Yat-Sen University, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]02-116-01
Record Dates: First submitted 2023-02-14; First posted 2023-02-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: interventions — camrelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined Therapy Using D-TACE, Gemcitabine and Cisplatin, and Camrelizumab (Experimental): D-TACE with cisplatin-eluting beads. More TACE can be done if clinically necessary.
  Camrelizumab (200 mg, Intravenous drips (ivd), D1/3W) plus Gem (1000 mg/m2, ivd, D1&8/3W) and Cis (25 mg/m2, ivd, D1&8/3W). Three weeks are one cycle of treatment. Chemotherapy lasted for no more than 12 cycles.
  Interventions: Drug: Camrelizumab; Drug: Gemcitabine Injection; Drug: Cisplatin injection; Drug: Cisplatin-Eluting Beads; Procedure: D-TACE

INTERVENTIONS:
Drug: Camrelizumab — 200mg on day1 of every 3 weeks, starting on day1 of cycle1
Drug: Gemcitabine Injection — 1000mg/m2 on day1 & day8 of every 3 weeks, starting on day1 of cycle 1
Drug: Cisplatin injection — 25mg/m2 on day1 & day8 of every 3 weeks, starting on day1 of cycle 1
Drug: Cisplatin-Eluting Beads — used for D-TACE
Procedure: D-TACE — TACE with Cisplatin-Eluting Beads (with Cis 30mg). More TACE can be done if clinically necessary.

SUMMARY:
The goal of this clinical trial is to learn about the combined therapy using drug-eluting bead-transarterial chemoembolization (D-TACE), gemcitabine (Gem) and cisplatin (Cis) chemotherapy, and PD-1 antibody in patients with advanced and unresectable intrahepatic cholangiocarcinoma (ICC). The main questions it aims to answer are:

* Whether combined therapy using D-TACE, Gem/Cis, and PD-1 works well to convert unresectable ICC to resectable.
* Whether combined therapy using D-TACE, Gem/Cis, and PD-1 is safe. Participants will receive D-TACE (CalliSpheres with Gem 30 mg), camrelizumab (200 mg) plus gemcitabine (1000 mg/m2) and cisplatin (25 mg/m2), and 24 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, male or female;
2. Histopathologically confirmed intrahepatic cholangiocarcinoma;
3. Tumor is unresectable assessed by the expert group (R0 resection CANNOT be achieved) and the life expectancy is more than 3 months;
4. Presence of at least one measurable lesion assessed using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST version 1.1);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Child-Pugh score ≤ 7;
7. Adequate organ function (neutrophil count of ≥1.5×10^9 cells/L, hemoglobin concentrations of ≥90 g/L, platelet cell count of ≥100×10^9 cells/L, bilirubin ≤1.5×ULN, Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 5×ULN, serum creatinine ≤ 1.5 x ULN, Thyroid stimulating hormone (TSH) ≤ 1 x ULN;
8. The patient must be required to sign an informed consent form;

Exclusion Criteria:

1. Patients who have received previous treatment with interventional therapy, radiotherapy, ablation, chemotherapy, targeted therapy, immunotherapy (PD-1, PD-L1, CLTA-4 antibody, etc), or surgery within the last 2 months;
2. Patients with other malignant tumors within the last 5 years, except for cured non-melanoma skin cancer, cervical carcinoma in situ, and papillary thyroid carcinoma;
3. Active tuberculosis infection. Patients with active tuberculosis infection within 1 year prior to enrollment; had a history of active tuberculosis infection more than 1 year before enrollment, did not receive formal anti-tuberculosis treatment or tuberculosis is still active;
4. Active infection requiring systemic therapy;
5. Human immunodeficiency virus (HIV) positive;
6. Have an active, known, or suspected autoimmune disease. Subjects who require only hormone replacement therapy for hypothyroidism and skin diseases that do not require systemic therapy may be enrolled;
7. Suffering from high blood pressure, and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
8. Abnormal blood coagulation (INR >1.5, or PT>ULN+4s, or APTT >1.5 x ULN), with a bleeding tendency or receiving thrombolytic or anticoagulant therapy;
9. Pregnant or lactating women;
10. Participated in other trials within the last 4 weeks;
11. Has a history of allergy to platinum;
12. Other factors that may influence the safety of the subject or the compliance of the test by the investigator. Serious illnesses (including mental illness), severe laboratory tests, or other family or social factors that require combined treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | 12 months
  Rate of unresectable ICC convert to resectable in combination therapy

SECONDARY OUTCOMES:
Incidence of adverse events | 12 months
  Rate of participants with treatment-related adverse events as assessed by CTCAE v4.0
Objective Response Rate (ORR) | 12 months
  ORR according to RECIST 1.1 using investigator assessment
Deepness of response (DpR) | 12 months
  DpR according to RECIST 1.1 using investigator assessment
Disease control rate (DCR) | 12 months
  DCR according to RECIST 1.1 using investigator assessment
Rate of R0 resection | 12 months
  R0 resection is defined as no tumor remains at the cutting edge and no tumor cells remain at the cutting edge under the microscope
Overall Survival (OS) | 12 months
  OS is defined as the time from date of combined theray start to the date of death from any cause or to the date of last follow-up if patients are alive.
Progression-free Survival (PFS) | 12 months
  From the beginning date of combined therapy to the date of disease progression. PFS according to RECIST 1.1 using investigator assessment
Recurrence-free Survival (RFS) | 12 months
  RFS is defined as the time between the date of surgery and the date of disease recurrence or death, whichever occurred first. RFS according to RECIST 1.1 using investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, MD&PhD, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No